CLINICAL TRIAL: NCT06815887
Title: Effect of Adding Magnesium Sulfate to Local Anesthetic in Combined Pectoral Nerve and Stellate Ganglion Block for Postoperative Pain Control After Modified Radical Mastectomy
Brief Title: Adding Magnesium Sulfate to Local Anesthetic in Combined Pectoral Nerve and Stellate Ganglion Block for Postoperative Pain Control After Modified Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Ali Ali, Specialist of Anesthesia, Intensive Care Unit and Pain Relief, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2311-201-091
Record Dates: First submitted 2025-02-01; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Magnesium Sulfate; Local Anesthetic; Pectoral Nerve; Stellate Ganglion Block; Postoperative Pain; Modified Radical Mastectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive the combined pectoralis nerve block II (PECS II)(20 mL) and stellate ganglion block (5 mL) using 0.5% bupivacaine (local anesthetic) without magnesium sulfate.
  Interventions: Drug: Bupivacaine
- Group B (Experimental): Patients will receive the combined (20 mL) pectoralis nerve block II (PECS II) and stellate ganglion block (5 mL) using 0.5% bupivacaine (local anesthetic) mixed with 2.5 mL magnesium sulfate (10%), i.e., 250 mg.
  Interventions: Drug: Bupivacaine + Magnesium sulfate

INTERVENTIONS:
Drug: Bupivacaine — Patients received the combined pectoralis nerve block II (PECS II) (20 mL) and stellate ganglion block (5 mL) using 0.5% bupivacaine (local anesthetic) without magnesium sulfate.
  Arms: Group A
Drug: Bupivacaine + Magnesium sulfate — Patients received the combined (20 mL) pectoralis nerve block II (PECS II) and stellate ganglion block (5 mL) using 0.5% bupivacaine (local anesthetic) mixed with 2.5 mL magnesium sulfate (10%), i.e., 250 mg.
  Arms: Group B

SUMMARY:
We aim to study the effect of adding magnesium sulfate as an adjuvant to the local anesthetic used in the combined Pectoralis Nerve Block II (PECS II) and stellate ganglion block for postoperative pain control in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
Post-operative pain from breast surgery can be controlled by regular pain medications such as paracetamol, non-steroidal anti-inflammatory (NSAIDs), and narcotics. Nerve blocks are commonly used as multimodal approaches for acute post-operative pain relief.

Pectoral and stellate ganglion blocks are regional anesthesia techniques that target the thoracic nerves and sympathetic nerve ganglia to provide analgesia for the upper extremity and chest regions. When combined, these blocks have shown promising results in alleviating perioperative pain for patients undergoing modified radical mastectomy.

Magnesium sulfate, a well-known adjuvant, has been studied extensively for its analgesic properties and anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Female gender.
* American Society of Anesthesiologists (ASA) physical status II or III.
* Patients scheduled for elective modified radical mastectomy for breast cancer.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.

Exclusion Criteria:

* Bleeding tendency due to coagulopathy,
* Patients with opioid dependence or alcohol or drug abuse,
* Significant liver and renal sufficiency
* Patients with psychiatric illnesses that prevent them from proper perception and assessment of pain.
* Local infection at the site of the block.
* Known hypersensitivity or allergy to magnesium sulfate or local anesthetics.
* Patients with chronic pain syndromes or pre-existing neuropathic pain conditions.
* Pregnant or lactating individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  With numeric rating scale (NRS) rest score ≥ 3 or NRS evoked score ≥ 4, morphine will be administered intravenously by a dose of 0.05 mg/kg at 30-minute intervals until NRS rest score < 3 or NRS evoked score < 4.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The severity of pain will be assessed postoperatively using a numeric rating scale (NRS) both at rest and evoked (0 = no pain and 10 = worst imaginable pain). NRS will be recorded at 1, 2, 4, 6, 8, 10, 12, and 24 hours postoperatively.
Time to first request analgesia | 24 hours postoperatively
  The time to first request analgesia will be recorded from the end of surgery till the first dose of morphine is administrated.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as nausea and vomiting will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of the study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.